CLINICAL TRIAL: NCT04517695
Title: Blood Volume, Components and Capillary Leak in ICU Patients With SARS-CoV-2 and Bacterial Infections
Brief Title: Blood Volume Assessment in COVID-19 and Bacterial Sepsis
Acronym: BVAC19
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-00896
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Acute Respiratory Distress Syndrome; Bacterial Sepsis; Bacterial Infections
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- COVID-19 ICU Patients: Patients who are admitted to the ICU with a confirmed SARS-CoV-2 infection
  Interventions: Device: BVA-100; Device: Transpulmonary Thermodilution (TPTD); Device: Sublingual Microcirculation
- ICU Patients with bacterial infection: Patients who are admitted to the ICU with a confirmed bacterial infection.
  Bacterial infection is defined as the clinical suspicion of a bacterial infection with the presence of two or more clinical markers of infection:
  * abnormal body temperature (>38C or <36C)
  * increased heart rate (>90 b/min),
  * increased respiratory rate > 20/min or a decreased arterial CO2: PaCO2 < 32 mmHg
  * Abnormal white blood cell count: < 4000 mm3 or > 12,000 /mm3 or > 10% immature cells
  OR
  * The presence of a positive (blood) culture with bacterial growth.
  Interventions: Device: BVA-100; Device: Transpulmonary Thermodilution (TPTD); Device: Sublingual Microcirculation

INTERVENTIONS:
Device: BVA-100 — The BVA-100 is a software package designed to calculate human blood volume using the method of tracer dilution. It uses tagged serum albumin.
Device: Transpulmonary Thermodilution (TPTD) — TPTD consists of placing a thermistor-equipped catheter in a central artery (usually the femoral or axillary artery) and injecting cold saline solution into a central vein through a central venous catheter.
  Other Names: PICCO
Device: Sublingual Microcirculation — With incident dark field imaging, the CytoCam device can record digital image sequences using a handheld camera. In the current study the camera will be used to non-invasively record images of the sublingual microcirculation.
  Other Names: CytoCam

SUMMARY:
In patients with SARS-CoV-2 or bacterial infection admitted to the intensive care unit (ICU), the state of the intravascular volume, the characteristics of the blood volume components, and the development of a vascular leak is currently unknown. The relationship of these parameters with parameters of cardiac performance, lung edema and sublingual microcirculatory perfusion parameters have never been studied.

DETAILED DESCRIPTION:
Acute respiratory failure related to infection by the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), is the main reason for ICU admission in in the majority of patients admitted to the ICU in this viral syndrome, and it presents a significant clinical challenge. Severe hypoxemia in these patients is thought to be related in part to generation of alveolar edema. This would be related to the specific infection related injury of the alveoli-capillary membrane, however other factors could be related to edema formation. Although patients meet criteria for the Acute Respiratory Distress Syndrome (ARDS), there is significant controversy about whether the lungs of the COVID-19 patients have the characteristics of ARDS and thus whether the treatment should mimic treatment of ARDS due to other causes. A general principle in ARDS patients is to avoid positive fluid balances as this may contribute to alveolar edema. Also, the guidelines on the management of COVID-19 patients by the Society of Critical Care Medicine advocate a conservative fluid strategy. However, uncorrected hypovolemia may result in additional organ dysfunction (especially kidney injury). The clinical fluid status is usually estimated by the presence of peripheral edema and daily fluid balances and thus prone to errors as these are poorly related to the circulating blood volume. Management of patients with sepsis based on blood volume measurements and red blood cell volume, to disclose true anemia, has been shown to improve outcome. Finally, the transudation of albumin in the extravascular space has been shown to be associated with outcome of critically ill patients. It is highly plausible that these parameters could help guide the care of COVID-19 patients given the available data in the literature, thus promoting better treatment of these patients.

This is a prospective multicenter study where the treatment team is blinded to the results of the study. The primary objective of the study is to describe the blood volume, the volume of blood components, the capillary leak and parameters of cardiac performance, lung edema and sublingual microcirculatory perfusion and their trajectory during the early phase of hospitalization of patients with SARS-CoV-2 or bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 or bacterial infection
* Patient admitted to the ICU
* Patient age is between 18 and 95 years
* Patent peripheral or central venous line from which blood draws can be made and through which the 131I bolus can be administered
* Arterial catheter considered indicated by primary team caring for the patient

Exclusion Criteria:

* Refused informed consent to participate in the study
* Pregnant or possible pregnant women
* Patient unlikely to survive more than 72h
* Patient with life sustaining treatment limitations (use of renal replacement therapy)
* Patient already on or likely to be placed on extra-corporeal membrane oxygenation support within 48h after admission
* Known allergy to iodine or iodinated 131I albumin
* Patients with chronic renal failure requiring renal replacement therapy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with a confirmed SARS-CoV-2 infection or bacterial infection
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Absolute Total Blood Volume | Day 1, Day of ICU Discharge (up to day 21)
  Absolute total blood volume calculated using BVA-100 software.
Change in Total Blood Volume Relative to Ideal Body Weight | Day 1, Day of ICU Discharge (up to day 21)
  Total blood volume relative to ideal body weight calculated using the BVA-100 software.
Change in Absolute Red Blood Cell Volume | Day 1, Day of ICU Discharge (up to day 21)
  Absolute red blood cell volume calculated using the BVA-100 software.
Change in Red Blood Cell Volume Relative to Ideal Body Weight | Day 1, Day of ICU Discharge (up to day 21)
  Red blood cell volume relative to ideal body weight calculated using the BVA-100 software.
Change in Absolute Plasma Volume | Day 1, Day of ICU Discharge (up to day 21)
  Absolute plasma volume calculated using the BVA-100 software.
Change in Plasma Volume Relative to Ideal Body Weight | Day 1, Day of ICU Discharge (up to day 21)
  Plasma volume relative to ideal body weight calculated using the BVA-100 software.
Change in Transudation Rate of Albumin | Day 1, Day of ICU Discharge (up to day 21)
  Transudation rate of albumin calculated using the BVA-100 software. An increase indicates the transudation rate increased during the observational period.
Change in Heart Rate | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. Heart rate expressed as beats per minute (BPM).
Change in Cardiac Output | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. Cardiac output expressed in liters per minute (L/min).
Change in Stroke Volume | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. Stroke volume expressed in milliliters per square meter (mL/m2).
Change in Systemic Vascular Resistance (SVR) | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. SVR expressed in dynes/second/cm^5.
Change in Global End Diastolic Volume (GEDV) Index | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. GEDV expressed in mL/m2.
Change in Intra-Thoracic Blood Volume Index (ITBVI) | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. ITBVI expressed in mL/m2.
Change in Extravascular Lung Water (EVLW) | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. EVLW expressed in mL/kg.
Maximum Stroke Volume | Up to Day of ICU Discharge (up to day 21)
  Measured using PICCO. Stroke volume expressed in mL/m2.
Minimum Stroke Volume | Up to Day of ICU Discharge (up to day 21)
  Measured using PICCO. Stroke volume expressed in mL/m2.
Maximum Pulse Pressure | Up to Day of ICU Discharge (up to day 21)
  Measured using PICCO. Pulse pressure expressed in millimeters of mercury (mmHg).
Minimum Pulse Pressure | Up to Day of ICU Discharge (up to day 21)
  Measured using PICCO. Pulse pressure expressed in millimeters of mercury (mmHg).
Change in Systolic Blood Pressure | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. Systolic blood pressure expressed in mmHg.
Change in Diastolic Blood Pressure | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. Diastolic blood pressure expressed in mmHg.
Mean Blood Pressure | Up to Day of ICU Discharge (up to day 21)
  Measured using PICCO. Blood pressure expressed in mmHg.
Change in Central Venous Pressure (CVP) | Day 1, Day of ICU Discharge (up to day 21)
  Measured using PICCO. CVP expressed in mmHg.

SECONDARY OUTCOMES:
Number of Participants with New Onset Renal Injury | Up to Day of ICU Discharge (up to day 21)
Number of Participants Requiring Renal Replacement Therapy | Up to Day of ICU Discharge (up to day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bakker, MD, PhD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - NYU Langone Health, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No